CLINICAL TRIAL: NCT01364285
Title: A Study of Patient Reported Outcomes After Stereotactic Radiosurgical Rhizotomy for Trigeminal Neuralgia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Soltys, Associate Professor of Radiation Oncology, Stanford University
Other Study IDs: SU-05252011-7808; IRB 16883 (Other: Stanford IRB)
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The investigators know little about how patients feel following radiosurgery treatment of trigeminal neuralgia. Patient satisfaction may ultimately be one of the most important outcome measures for an individual patient; however, this has not been adequately assessed or followed. Multiple questions remain unanswered, including whether there is a correlation between patient satisfaction, the level of their current pain score, and the presence and degree of facial numbness, a possible side effect after radiosurgery. Therefore, the goal of this study is to gather this information from the patients who received radiosurgery for trigeminal neuralgia at Stanford and evaluate post-treatment patient satisfaction, the degree of facial numbness, and current pain score. This data will help the investigators understand outcomes that are important for patient satisfaction following treatment of a chronic pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All of the patients since 2000 who have undergone stereotactic radiosurgical rhizotomy at Stanford for treatment of trigeminal neuralgia.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the patients since 2000 who have undergone stereotactic radiosurgical rhizotomy at Stanford for treatment of trigeminal neuralgia.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction following CyberKnife radiosurgery | 1 year
  To assess patient reported outcomes following stereotactic radiosurgical rhizotomy for trigeminal neuralgia.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Choi, Principal Investigator — Stanford University; Scott Soltys, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States